CLINICAL TRIAL: NCT02594371
Title: An Open-Label, Randomized, Multicenter, Phase 3 Study to Determine the Safety, Tolerability, and Tumor Response of Oraxol and Its Comparability to IV Taxol or Generic IV Paclitaxel in Subjects With Metastatic Breast Cancer
Brief Title: Ph3 Study To Determine Safety,Tolerability&Tumor Response Of Oraxol Compared To Taxol In Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORAX-001
Record Dates: First submitted 2015-10-28; First posted 2015-11-03 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oraxol (paclitaxel + HM30181AK-US) (Experimental): Oraxol paclitaxel - supplied as 30-mg capsules
  Oraxol HM30181 methansulfonate monohydrate - supplied as 15-mg HM30181AK-US tablets
  Interventions: Drug: Oraxol
- IV paclitaxel (Active Comparator): IV paclitaxel - supplied as Taxol or generic
  Interventions: Drug: IV paclitaxel

INTERVENTIONS:
Drug: Oraxol
  Other Names: HM30181 methanesulfonate monohydrate; Oral paclitaxel capsules
  Arms: Oraxol (paclitaxel + HM30181AK-US)
Drug: IV paclitaxel
  Arms: IV paclitaxel

SUMMARY:
To determine the safety and tolerability of Oraxol as compared to IV paclitaxel in metastatic breast cancer

DETAILED DESCRIPTION:
This is a Phase 3, open-label, randomized, multicenter study in approximately 360 adult female subjects with histologically- or cytologically-confirmed breast cancer that is metastatic for whom treatment with IV paclitaxel monotherapy has been recommended by their oncologist. Approximately 400 subjects will be enrolled to provide 360 evaluable subjects. The subjects must have measurable metastatic target lesion disease as per RECIST v1.1 criteria. Subjects will be randomized in a 2:1 ratio to either Oraxol or IV paclitaxel (as Taxol or generic).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Women ≥18 years of age
3. Histologically- or cytologically-confirmed breast cancer for whom IV paclitaxel (as Taxol or generic) monotherapy has been recommended by their oncologist
4. Measurable metastatic target lesion disease measurable by CT scan as per RECIST v1.1 criteria
5. Adequate hematological status as demonstrated by not requiring granulocyte-colony stimulating factor (G-CSF) or transfusion support to achieve the following at Screening:

   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelet count ≥100 x 109/L
   * Hemoglobin ≥10 g/dL
6. Adequate liver function as demonstrated by:

   * Total bilirubin within normal limits (WNL)
   * Alanine aminotransferase and aspartate aminotransferase ≤3 x upper limit of normal (ULN)
   * Alkaline phosphatase ≤3 x ULN or ≤5 x ULN if bone metastasis is present
   * Gamma glutamyl transferase (GGT) ≤5 x ULN
7. Adequate renal function as demonstrated by serum creatinine ≤1.5 x ULN
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
9. Life expectancy of at least 6 months, in the judgement of the investigator
10. Subjects must be postmenopausal (≥12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or must be using effective contraception and agree to used of contraception for 30 days after their last dose of assigned study treatment.
11. Subjects who are of childbearing potential must have a negative screening serum pregnancy test.

Exclusion Criteria:

1. Have not recovered to ≤ Grade 1 toxicity from previous anticancer treatments or previous investigational products
2. If previously treated with a taxane (paclitaxel or docetaxel) as part of anthracycline-based adjuvant chemotherapy or for metastatic disease, the subject relapsed less than 1 year following treatment
3. Only evidence of metastatic disease is to bone or other nontarget or nonmeasurable lesions (including, for example, ascites or plural effusion) according to RECIST v1.1 criteria
4. Central nervous system metastasis, including leptomeningeal involvement
5. Received IPs within 14 days or 5 half-lives of the first study dosing day, whichever is longer
6. Are currently receiving other medications intended for the treatment of their malignancy
7. Received radiation therapy within 2 weeks prior to signing informed consent and those for whom radiation therapy is planned within 6 months from the time of signing informed consent
8. Women who are pregnant or breastfeeding
9. Taking a medication known to be a strong P-gp inhibitor or inducer within 14 days of starting treatment
10. Taking an oral medication with a narrow therapeutic index known to be a P-gp substrate within 24 hours prior to start of treatment
11. Taking a medication known to be a strong cytochrome P450 (CYP) 3A4 inhibitor (eg, ketoconazole) or inducer (eg, rifampin or St. John's Wort) within 14 days of starting treatment
12. Taking a medication known to be a strong inhibitor (eg, gemfibrozil) or inducer (eg, rifampin) of CYP2C8 within 14 days of starting treatment
13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myocardial infarction within the last 6 months, unstable angina pectoris, cardiac arrhythmia, chronic pulmonary disease requiring oxygen, known bleeding disorders, or any concomitant illness or social situation that would limit compliance with study requirements
14. Major surgery to the upper GI tract, or have a history of GI disease or other medical condition that, in the opinion of the Investigator may interfere with oral drug absorption
15. History of significant hypersensitivity-type reactions to paclitaxel or Cremophor EL (polyoxyl 35 castor oil, NF) that would contraindicate the use of IV paclitaxel formulated with Cremophor EL
16. Known allergic reaction or intolerance to contrast media
17. Documented history of true systemic allergic reaction to 3 or more medications
18. For whom the Investigator believes that participation in this study would not be acceptable
19. Known chronic hepatitis or cirrhosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Tumor response as determined by response criteria | 19 to 22 weeks
  Tumor response is evaluated using the response evaluation criteria in solid tumors (RECIST v1.1 criteria).
Safety and tolerability assessments of Oraxol compared with IV paclitaxel, as determined by laboratory, adverse event (AE) and serious adverse event (SAE) information | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to ~48 months (expected end of study).]
  Safety assessments will consist of determining and recording all AEs and SAEs; laboratory evaluation of hematology, blood chemistry, and urine analyses; periodic measurement of vital signs and electrocardiograms (ECGs); and the performance of physical examinations, as detailed in the schedule of procedures and assessments of the protocol

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to ~48 months (expected end of study).
  The endpoint of progression-free survival is defined as not having died or progression of disease. Lost to follow-up will be considered as censored.
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to ~48 months (expected end of study).
  The endpoint of overall survival is defined as death, confirmed alive, and lost to follow-up. Alive and lost to follow-up will be considered as censored.

CONTACTS AND LOCATIONS:
Overall Officials: David Cutler, MD, Study Director — Kinex Pharmaceuticals Inc.
Locations (45):
- Argentina (15):
  - Centro de Investigacion Pergamino SA, Pergamino, Buenos Aires
  - Clinica Universitaria Privada Reina Fabiola, Córdoba, Córdoba Province
  - IONC, Córdoba, Córdoba Province
  - Centro Oncologico Infinito, Santa Rosa, La Pampa Province
  - Fundación Koriza, Santa Rosa, La Pampa Province
  - Clinica Viedma, Viedma, Río Negro Province
  - CEMEDIC, Buenos Aires
  - COIBA, Buenos Aires
  - Fundación Investigar, Buenos Aires
  - Fundación Centro Oncológico Riojano Integral (CORI), La Rioja
  - CAIPO, San Miguel de Tucumán
  - Centro Medico San Roque, San Miguel de Tucumán
  - Hospital Provincial del Centenario, Santa Fe
  - Instituto de Oncologia de Rosario, Santa Fe
  - Sanatorio Britanico, Santa Fe
- Chile (5):
  - Fundación Arturo López Pérez, Santiago
  - Hospital de Referencia de Salud Cordillera Unidad de Patología Mamaria, Santiago
  - Hospital San Borja Arriarán, Santiago
  - IRAM, Santiago
  - Clínica Alemana Temuco, Temuco
- Colombia (4):
  - Instituto Nacional de Cancerología E.S.E., Bogotá
  - Fundación Colombiana de Cancerología Clinica Vida, Medellín
  - Fundación Hospitalaria San Vicente de Paúl, Medellín
  - Hemato Oncologos S.A., Valle
- Dominican Republic (3):
  - Hospital Metropolitano de Santiago (HOMS), Santiago de los Caballeros
  - Clinical Research, Santo Domingo
  - Hospital General de la Plaza de la Salud, Santo Domingo
- Ecuador (3):
  - Hospital SOLCA, Guayaquil
  - Hospital Carlos Andrade Martín, Quito
  - Hospital SOLCA, Quito
- El Salvador (2):
  - Espemedic, San Salvador
  - Hospital Diagnotico Clinica Oncologica & Cancer Research, San Salvador
- Guatemala (7):
  - American Cancer Center, Guatemala City
  - CELAN Clínica Médica, Guatemala City
  - Clinica Privada, Guatemala City
  - Clínica Privada, Guatemala City
  - Grupo Angeles, S.A., Guatemala City
  - Oncomedica en Guatemala, Guatemala City
  - CRESEM, Quetzaltenango
- Honduras (2):
  - Excel Medica, Cortés
  - Tecnología en Investigación, Cortés
- Centro Hemato Oncológico Panamá, Panama City, Panama
- Peru (3):
  - Clínica Oncológica Miraflores, Lima
  - Hospital Cayetano Heredia, Lima
  - Hospital Nacional del Arzobispo Loayza, Lima

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rugo HS, Umanzor GA, Barrios FJ, Vasallo RH, Chivalan MA, Bejarano S, Ramirez JR, Fein L, Kowalyszyn RD, Kramer ED, Wang H, Kwan MR, Cutler DL; Oraxol Study Consortium Investigators. Open-Label, Randomized, Multicenter, Phase III Study Comparing Oral Paclitaxel Plus Encequidar Versus Intravenous Paclitaxel in Patients With Metastatic Breast Cancer. J Clin Oncol. 2023 Jan 1;41(1):65-74. doi: 10.1200/JCO.21.02953. Epub 2022 Jul 20. PMID 35858154